CLINICAL TRIAL: NCT01650415
Title: Random Control Trial to Evaluate the Safety and Efficacy of Erythropoietin Therapy for Children With Cerebral Palsy -Patient, Principle Investigator, Observer Blind
Brief Title: Erythropoietin Therapy for Children With Cerebral Palsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bundang CHA Hospital (Other)
Collaborators: LG Life Sciences (Industry)
Responsible Party: Principal Investigator, MinYoung Kim, M.D., Associate Professor, Bundang CHA Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPEPO
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Erythropoietin; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy | interventions — Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erythropoietin and Rehabilitation (Experimental): recombinant human erythropoietin injection and active rehabilitation
  Interventions: Drug: Erythropoietin
- Placebo and Rehabilitation (Placebo Comparator): Placebo erythropoietin and rehabilitation
  Interventions: Drug: Placebo erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — twice a week for 1 month
  Other Names: Espogen
  Arms: Erythropoietin and Rehabilitation
Drug: Placebo erythropoietin — twice a week for 1 month
  Arms: Placebo and Rehabilitation

SUMMARY:
This randomized placebo-controlled trial aims to investigate the efficacy and safety of erythropoetin for children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy is a disorder of movement and posture resulted from a nonprogressive lesion or injury of the immature brain. It is a leading cause of childhood onset disability.

Many experimental animal studies have revealed that erythropoietin is useful to repair neurological injury in brain. The main mechanism of erythropoietin is supposed as follows;

1. Neuroprotection effect
2. Angiogenesis
3. Anti-inflammation.

On the basis of many experimental studies, erythropoietin is suggested as a therapeutic method for cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy
* Abnormal Muscle Tone
* Abnormal Brain MRI
* Willing to Comply with All Study Procedure

Exclusion Criteria:

* Known Genetic Disorder
* Other Etiologies Contributing Developmental Delay
* Coagulopathy
* Initial high Erythropoietin level in Serum
* Previous Erythropoietin Treatment before 3 months
* Presence of Drug Hypersensitivity Related to the Study Remedy
* Intractable Seizure Disorder
* Poor Cooperation of Guardian including Inactive Attitude for Rehabilitation

Ages: 4 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in Quality of Movement | Baseline - 2 months
  GMPM (Gross Motor Performance Measure) as a standardized measurement tool for assessing quality of movement regarding 3 properties of 5 ones: alignment, coordination, dissociated movement, stability, and weight shift. The interrater reliability of GMPM subscores and total scores was 0.758-0.886 (subject n=75, tester n=10).

SECONDARY OUTCOMES:
Changes in Gross Motor Function | Baseline - 2 months
  GMFM (Gross Motor Function Measure) as a standardized measurement tool for assessing Gross Motor Function consisting of 6 sub-scales; lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping. The measured interrater reliability of GMFM subscores and total scores was 0.974 - 0.997 (subject n=101, tester n=10) and intrarater reliability of GMFM subscores and total scores between one most experienced rater and another newly t rained rater was 0.994 - 1.000 (subject n=101, tester n=2).
Changes in Neurodevelopmental Outcomes | Baseline - 2 months
  K-BSID-II (Korean version of Bayley Scale of Infant Development-II) Motor and Mental Scales. The measured intrarater and interrater reliability of K-BSID-II motor and mental scales was 0.92 - 0.99 (subject n=55, tester n=10).
Changes in Motor Development | Baseline - 2 months
  AIMS (Alberta Infant Motor Scale)to measure the motor development
Changes in Spasticity | Baseline - 2 months
  MAS (modified Ashworth Scale)measured at biceps, hip adductor, hamstring, heel cord

CONTACTS AND LOCATIONS:
Overall Officials: Minyoung Kim, M.D., Ph.D., Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea